CLINICAL TRIAL: NCT05163184
Title: Physiologic Tension of the Abdominal Wall
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rosen, Professor of Surgery, The Cleveland Clinic
Other Study IDs: 21-1036
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Abdominal Wall Hernia
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparotomy: Patients undergoing laparotomy

SUMMARY:
Restoring the physiologic tension of the abdominal wall is a key concept in abdominal wall reconstruction. Yet little is known quantitatively about the normal tension of the abdominal wall. To better understand the ideal tension for abdominal wall reconstruction, the physiologic tension of the abdominal wall needs to be measured. This study aims to measure the tension of the abdominal wall during laparotomy closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparotomy
* Patient able to provide informed consent

Exclusion Criteria:

* Presence of a ventral hernia
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing laparotomy without a ventral hernia.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Abdominal wall tension at laparotomy | Tension measurements will be recorded immediately. No further data collection or patient follow-up will occur postoperatively.
  The tension necessary to bring the abdominal wall to the midline during laparotomy will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No